CLINICAL TRIAL: NCT04073992
Title: Chronic Insomnia and CSF Markers of Dementia - Effects of Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 833798
Record Dates: First submitted 2019-08-27; First posted 2019-08-29 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Insomnia Chronic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive behavioral treatment of insomnia (CBT-I) (Experimental): Eight weeks of cognitive behavioral treatment of insomnia.
  Interventions: Behavioral: cognitive behavioral treatment of insomnia

INTERVENTIONS:
Behavioral: cognitive behavioral treatment of insomnia — A behavioral modification program consisting of 8 clinic sessions focused on sleep hygiene, stimulus control, sleep restriction, and cognitive restructuring.

SUMMARY:
The longstanding view has been that insomnia, and other forms of sleep disturbance, emerge as a consequence of dementia and are the result of progressive neuronal damage. However, there is growing evidence that the direction of causation may go both ways, with sleep disturbance potentially increasing vulnerability to dementia. Longitudinal studies have found that sleep disturbance often precedes and increases risk for dementia by several years. The purpose of this study is to examine whether treatment of insomnia with cognitive behavioral therapy (CBT-I) is associated with a decrease in dementia biomarkers found in cerebrospinal fluid (CSF). Fifteen adults age 30-50 with chronic insomnia will undergo overnight polysomnography and CSF sampling in the morning. This will be followed by 8 weeks of treatment with CBT-I and then repeat CSF sampling.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-50
* Men and women
* Meet DSM5 Diagnostic Criteria for insomnia disorder

Exclusion Criteria:

* Diagnosis or evidence of sleep disorders other than insomnia as determined by the screening questionnaires and clinical history
* Women who have been pregnant or lactating within the past six months
* Non-fluency in spoken or written English
* Current or past month shiftwork defined as working during the evening or night shift
* Current use of medications or OTC products that impact sleep
* Evidence of neurological abnormalities that could include the risks associated with lumbar puncture (e.g.papilledema, mass lesion, Chiari malformation).

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
CSF markers related to dementia | 8 weeks
  CSF levels of the proteins tau and beta amyloid

CONTACTS AND LOCATIONS:
Overall Officials: Philip Gehrman, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No